CLINICAL TRIAL: NCT02349997
Title: The First Affiliated Hospital of Nanjing Medical University
Brief Title: Fluid Shift on Obstructive and Central Sleep Apnea
Status: Completed | Type: Observational
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Ning Ding, Department of Respiratory Medicine, The First Affiliated Hospital of Nanjing Medical University, Nanjing Medical University
Other Study IDs: 2014-SR-168
Record Dates: First submitted 2015-01-18; First posted 2015-01-29 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Apnea (Central and Obstructive)
Keywords: central sleep apnea; Cheyne-Stokes respiration; obstructive sleep apnea; chronic heart failure; fluid shift
MeSH Terms: conditions — Apnea; Sleep Apnea, Central; Cheyne-Stokes Respiration; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- OSA group: Of the 180 heart failure patients,20 OSA were enrolled. Clinical evaluations including NYHA class, electrocardiographic, echocardiographic, arterial blood gas analysis findings, baseline medication, and 6-minute walk test (6MWT) were recorded.
  The fluid index, head and neck CT and pharyngeal resistance were tested at 20:00. Then a full night PSG and percutaneous PaCO2 were performed. The fluid index, head and neck CT and pharyngeal resistance were repeated at 6:00 after PSG.
  The volume of fluid shift from legs to head and neck,inside diameter of the upper airway, and water content of neck soft tissue were calculated. The lung-to-finger circulation time and loop gain were measured.
  Interventions: Other: no interventions
- CSA group: Of the 180 heart failure patients,20 CSA were enrolled. Clinical evaluations including NYHA class, electrocardiographic, echocardiographic, arterial blood gas analysis findings, baseline medication, and 6-minute walk test (6MWT) were recorded.
  The fluid index, head and neck CT and pharyngeal resistance were tested at 20:00. Then a full night PSG and percutaneous PaCO2 were performed. The fluid index, head and neck CT and pharyngeal resistance were repeated at 6:00 after PSG.
  The volume of fluid shift from legs to head and neck,inside diameter of the upper airway, and water content of neck soft tissue were calculated. The lung-to-finger circulation time and loop gain were measured.
  Interventions: Other: no interventions

INTERVENTIONS:
Other: no interventions — This is an observational study and no intervention applied.

SUMMARY:
Fluid retention in the legs due to chronic heart failure (CHF) during the daytime may redistribute to neck when with supine positioning at night. A portion of the shifted fluid accumulates in the neck, and narrows the upper airway, predisposing the patient to obstructive sleep apnea (OSA) and central sleep apnea (CSA). However, the mechanism of overnight fluid shift on OSA and CSA remains unclear. The investigators pre-experiment demonstrated there may be a different mechanism of overnight fluid shift on OSA and CSA. The accumulation of water content in neck soft tissue increases neck circumference and leads to pharyngeal resistance, upper airway collapse and causes OSA. The effect of nocturnal fluid shift on CSA may be because of increasing of chemosensitivity (fluctuation of PaCO2), circulation delay and hemodynamic disordered. This study is aimed to explore the different mechanism of overnight fluid shift on OSA and CSA by comparing the changes of upper airway (inside diameter, water content, and pharyngeal resistance), PaCO2, circulation delay (lung-to-finger circulation time) and hemodynamic (loop gain).

DETAILED DESCRIPTION:
Methods:

Between June 2015 and December 2017, 180 patients with chronic heart failure caused by rheumatic heart disease, cardiomyopathy and coronary heart disease (in Cardiology Department and Cardiothoracic Surgery Department of the First Affiliated Hospital of Nanjing Medical University), were screened for sleep apnea by polysomnography (PSG). Of them, 20 obstructive sleep apnea (OSA) and 20 central sleep apnea (CSA) were enrolled. Clinical evaluations including NYHA class, electrocardiographic, echocardiographic, arterial blood gas analysis findings, baseline medication, and 6-minute walk test (6MWT) were recorded.

The fluid index, head and neck CT and pharyngeal resistance were tested at 20:00. Then a full night PSG and percutaneous PaCO2 were performed. The fluid index, head and neck CT and pharyngeal resistance were repeated at 6:00 after PSG.

The volume of fluid shift from legs to head and neck,inside diameter of the upper airway, and water content of neck soft tissue were calculated. The lung-to-finger circulation time and loop gain were measured.

1. Mechanism of overnight fluid shift on OSA:

   Fluid shift volume from legs to head and neck,inside diameter of upper airway, water content of neck soft tissue, percutaneous PaCO2, severity of sleep apnea, minimum SP02, lung-to-finger calculation time and loop gain were measured at 22:00 and repeated at 6:00 next morning in patients with OSA.Correlations between changes of fluid shift volume and changes in diameter of upper airway, water content of neck soft tissue, PaCO2, minimum SP02, lung-to-finger calculation time and loop gain were analyzed.
2. Mechanism of overnight fluid shift on CSA:

Fluid shift volume from legs to head and neck,inside diameter of upper airway, water content of neck soft tissue, percutaneous PaCO2, severity of sleep apnea, minimum SP02, lung-to-finger calculation time and loop gain were measured at 22:00 and repeated at 6:00 next morning in patients with CSA.Correlations between changes of fluid shift volume and changes in diameter of upper airway, water content of neck soft tissue, PaCO2, minimum SP02, lung-to-finger calculation time and loop gain were analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. patients with chronic heart failure caused by rheumatic heart disease, cardiomyopathy and coronary heart disease
2. aged between 18 to 70 years
3. with symptomatic stable heart failure, New York Heart Association (NYHA) class >= II despite optimal drug therapy
4. patients combined with sleep apnea (apnea-hypopnea index >=10/h) according to the results of polysomnograph.

Exclusion Criteria:

1. history of stroke or clinical signs of peripheral or central nervous system disorders
2. chronic obstructive pulmonary disease or history of asthma
3. enrolment in another clinical study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with chronic heart failure caused by rheumatic heart disease, cardiomyopathy and coronary heart disease.
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2015-01; Primary Completion 2018-12-31 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
nocturnal fluid shift, as determined by change in leg fluid volume | up to 24 months
  Nocturnal fluid shift was measured for 40 enrolled participants.
pharyngeal resistance,as the change from baseline in pharyngeal air-flow resistance | up to 24 months
  Pharyngeal resistance was measured for 40 enrolled participants.
Lung to Finger Circulation Time | up to 24 months
  Lung to Finger Circulation Time was measured for 40 enrolled participants.
Loop Gain | up to 24 months
  Loop Gain was measured for 40 enrolled participants
apnea-hypopnea index, as the severity of sleep apnea. | up to 24 months
  Apnea-hypopnea index was measured for 40 enrolled participants.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Yumino D, Redolfi S, Ruttanaumpawan P, Su MC, Smith S, Newton GE, Mak S, Bradley TD. Nocturnal rostral fluid shift: a unifying concept for the pathogenesis of obstructive and central sleep apnea in men with heart failure. Circulation. 2010 Apr 13;121(14):1598-605. doi: 10.1161/CIRCULATIONAHA.109.902452. Epub 2010 Mar 29. PMID 20351237
- [Background] Ding N, Lin W, Zhang XL, Ding WX, Gu B, Ni BQ, Zhang W, Zhang SJ, Wang H. Overnight fluid shifts in subjects with and without obstructive sleep apnea. J Thorac Dis. 2014 Dec;6(12):1736-41. doi: 10.3978/j.issn.2072-1439.2014.11.19. PMID 25589967
- [Background] Kasai T, Motwani SS, Elias RM, Gabriel JM, Taranto Montemurro L, Yanagisawa N, Spiller N, Paul N, Bradley TD. Influence of rostral fluid shift on upper airway size and mucosal water content. J Clin Sleep Med. 2014 Oct 15;10(10):1069-74. doi: 10.5664/jcsm.4102. PMID 25317087